CLINICAL TRIAL: NCT06726889
Title: Optimizing an Intervention to Increase Oral Medication Adherence for Metastatic Breast Cancer Patients
Brief Title: Increasing Oral Medication Adherence for Metastatic Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 2014
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Metastatic Breast Cancer; Oral Anticancer Agents; Oral Medication Adherence
MeSH Terms: conditions — Breast Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Standard Care + DSS + Reminders + Feedback: Patients will receive educational material through a web-page, personalized reminders and feedback messages by physician
  Interventions: Behavioral: Standard care; Behavioral: Decision Support System (DSS); Behavioral: Reminders; Behavioral: Feedback
- Standard Care + DSS + Reminders: Patients will receive educational material through a web-page and personalized reminders
  Interventions: Behavioral: Standard care; Behavioral: Decision Support System (DSS); Behavioral: Reminders
- Standard Care + DSS + Feedback: Patients will receive educational material through a web-page and feedback messages by physician
  Interventions: Behavioral: Standard care; Behavioral: Decision Support System (DSS); Behavioral: Feedback
- Standard Care + DSS: Patients will receive educational material through a web-page
  Interventions: Behavioral: Standard care; Behavioral: Decision Support System (DSS)
- Standard Care + Reminders + Feedback: Patients will receive personalized reminders and feedback messages by physician
  Interventions: Behavioral: Standard care; Behavioral: Reminders; Behavioral: Feedback
- Standard Care + Reminders: Patients will receive personalized reminders
  Interventions: Behavioral: Standard care; Behavioral: Reminders
- Standard Care + Feedback: Patients will receive feedback messages by physician
  Interventions: Behavioral: Standard care; Behavioral: Feedback
- Standard Care: Patient will not receive any additional interventions
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Standard care — Patient will not receive any additional interventions
Behavioral: Decision Support System (DSS) — DSS will be used to deliver educational material through a web-page (in Italian language) accessible through a link
  Groups: Standard Care + DSS; Standard Care + DSS + Feedback; Standard Care + DSS + Reminders; Standard Care + DSS + Reminders + Feedback
Behavioral: Reminders — Personalized reminders will be delivered to patients through a common messaging application (WhatsApp)
  Groups: Standard Care + DSS + Reminders; Standard Care + DSS + Reminders + Feedback; Standard Care + Reminders; Standard Care + Reminders + Feedback
Behavioral: Feedback — Feedback message will be delivered by physician to patients, through WhatsApp, after medication diary revision
  Groups: Standard Care + DSS + Feedback; Standard Care + DSS + Reminders + Feedback; Standard Care + Feedback; Standard Care + Reminders + Feedback

SUMMARY:
Aim of this study is to optimize an adherence increasing intervention designed for metastatic Breast Cancer (BC) patients by applying a full factorial design in order to evaluate the optimal combination of three different intervention components.

DETAILED DESCRIPTION:
Today different types of Oral Anticancer Agents (OAA) are commonly prescribed to Breast Cancer (BC) patients. Patients are reported to prefer the oral modality of administration over the intravenous one for its convenience, flexibility, and easier assumption; nonetheless, the phenomenon of medication non-adherence is well-documented.

Although several interventions have been designed and tested in order to foster medication adherence among BC patients, the great majority of them were focused on adherence to endocrine therapy for early-stage BC patients, with only few exceptions involving metastatic BC patients or considering adherence to other types of OAA.

The aim of this work is to optimize an adherence increasing intervention designed for metastatic BC patients. This will be achieved by applying a full factorial design in order to evaluate the optimal combination of three different intervention components (informative documentation, personalized reminders and feedback).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of metastatic BC
* Patients with a prescription for any OAA (i.e. oral chemotherapy, endocrine therapy, and Cyclin-Dependent Kinase 4/6 Inhibitors)
* Age >18 years old
* Patients with a personal smart phone with internet access
* Willingness and ability to comply with scheduled visits and other trial procedures
* Understanding and speaking Italian language
* Written informed consent

Exclusion Criteria:

* Psychiatric disorders or conditions that might impair the ability to give informed consent
* Comorbidity that may impact on compliance to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic breast cancer patients with a prescription for any Oral Anticancer Agent
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Adherence to oral medication | 7 months
  Adherence rates will be evaluated as the percentage of doses correctly assumed compared to the total prescribed

SECONDARY OUTCOMES:
Depressive symptoms evaluation | 7 months
  Collection of Beck Depression Inventory II (BDI-II) questionnaire (minimum value: 0, maximum value: 3 - higher scores mean greater depression)
Anxiety evaluation | 7 months
  Collection of State-Trait Anxiety Inventory (STAI) questionnaire (minimum value: 1, maximum value: 4 - higher scores signify greater anxiety)
Quality of life evaluation | 7 months
  Completion of European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) EORTC-QLQ-C30 (minimum value: 1, maximum value: 4 - higher scores mean a greater agreement with the statement)
Health-related quality of life evaluation | 7 months
  Completion of European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality of Life Questionnaire (EORTC-QLQ-BR23) (minimum value: 1, maximum value: 4 - higher scores mean a greater agreement with the statement)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravettoni, MD, Principal Investigator — European Istitute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy